CLINICAL TRIAL: NCT04047732
Title: A Phase I/II Clinical Trial of Topical KB105, a Replication-incompetent, Non-integrating HSV-1 Vector Expressing Human Transglutaminase 1 (TGM1) for the Treatment of TGM1-deficient Autosomal Recessive Congenital Ichthyosis (ARCI)
Brief Title: Topical KB105 Gene Therapy for the Treatment of TGM1-deficient Autosomal Recessive Congenital Ichthyosis (ARCI)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB105-001
Record Dates: First submitted 2019-07-29; First posted 2019-08-07 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: TGM-1 Related Autosomal Recessive Congenital Ichthyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topical KB105 (Experimental): HSV1-TGM1 vector (KB105)
  Interventions: Biological: KB105

INTERVENTIONS:
Biological: KB105 — KB105, a replication-incompetent, non-integrating HSV-1 vector expressing human transglutaminase 1 (TGM1) formulated as a topical gel
  Other Names: HSV1-TGM1

SUMMARY:
This study is an intra-patient comparison of KB105 and placebo-administered Target Areas. The primary objectives of this study are to evaluate safety and Investigator Global Assessment (IGA) scale improvement of topically administered KB105.

DETAILED DESCRIPTION:
Up to six adult subjects are planned for the Phase I portion of this study. Subjects are enrolled upon obtaining consent and meeting entry criteria. This study is an intra-patient comparison of KB105 and placebo-administered Target Areas. Patients will be evaluated for safety, and Target Areas will be assessed individually with the IGA and VIIS scales. Target Areas will be imaged and evaluated for safety and efficacy. Subjects will be on-trial for approximately 3.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of TGM1-deficient ARCI with a null TGM-1 mutation;
* Clinical diagnosis of lamellar ichthyosis;
* Age: 18 years old or older;
* Individual site IGA score of 3 to 4 at the target areas
* Subject is, in the opinion of the Investigator, able to understand thestudy, cooperate with the study procedures, and is willing to return to the clinic for all required follow-up visits;
* Except for their moderate-to-severe ARCI, subject is in good general health; and
* Willing and able to give consent/assent.

Exclusion Criteria:

* Medical instability limiting ability to travel to the investigative center;
* Medical illness expected to complicate participation, such as an active infection with: HIV, hepatitis B (as determined by hepatitis B surface antigen screening), hepatitis C (as determined by detection of hepatitis C antibodies or a positive result of hepatitis C);
* Patient has a physical condition or other dermatological disorder (e.g., atopic, seborrheic, or contact dermatitis, psoriasis, tinea infections, etc.) which, in the Investigator's opinion, might impair evaluation of the Target Areas or which exposes the patient to unacceptable risk by study participation;
* Pregnant or breast-feeding women, or women planning to become pregnant or to breast-feed. Women of childbearing potential must have a negative urine pregnancy test at the Screening visit and Day 1 visit and must commit to using an acceptable form of contraception during the entire study period, up to three months after last KB105 administration. Women using oral contraception must also have done so for 3 months prior to Baseline or will be willing to use a combination of barrier methods. To be considered not of childbearing potential, women must be post-menopausal for at least 1 year or surgically sterile
* Known allergy to any of the constituents of the product
* Hypersensitivity to local anesthesia (e.g., lidocaine/prilocainecream)
* Current enrollment in a clinical trial
* Treatment with an investigational drug or investigational device within 30 days prior to Day 1
* Male who is not surgically sterile nor willing to use effective forms of contraception from Day 1 until 3 months following the last dose of study drug.
* Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 12 weeks
  Incidence of treatment-emergent adverse events
Investigator's Global Assessment (IGA) of disease severity | Up to 12 weeks
  Improvement of disease severity in the treatment area assessment through Investigator's Global Assessment (IGA)

SECONDARY OUTCOMES:
Visual Index for Ichthyosis Severity (VIIS) scale, lamellar (L) standard | Up to 12 weeks
  Improvement of disease severity in the treatment area through use of the Visual Index for Ichthyosis Severity scale, lamellar (VIIS-L) standard assessment. The VIIS-L is a 4-point visual scale with 1 representing normal skin and 5 representing severe ichthyosis.
Immunofluorescence microscopy | Up to 12 weeks
  Level of transglutaminase 1 in KB105-administered skin as measured by immunofluorescence microscopy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No